CLINICAL TRIAL: NCT06272318
Title: Vital Signs Blood Pressure Trial
Status: Not yet recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David R. Drover, Principal Investigator, Stanford University
Other Study IDs: 74131
Record Dates: First submitted 2024-02-06; First posted 2024-02-22 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases; Hypertension; Blood Pressure
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension | interventions — serglycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood Pressure Cuff, EKG, PPG — A blood pressure cuff, an EKG, and a PPG will be utilized to collect subject vitals.

SUMMARY:
The purpose of this study is collect subject vitals with a blood pressure cuff, electrocardiogram (ECG), and photoplethysmogram (PPG). This data can then be used to develop a reliable, accurate, noninvasive, and continuous blood pressure monitoring device.

ELIGIBILITY:
Inclusion Criteria:

* Age >17 and <65 years
* BMI >20 and <35

Exclusion Criteria:

* Age <18 or >64
* BMI <20 or >35
* Pregnancy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants with a range of health conditions are needed for this study, including those with cardiac or blood pressure issues, as well as individuals who are considered healthy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Collection of Subject Name (optional) | Less than 1 minute
Collection of Subject Height | Less than 1 minute
  Height in meters
Collection of Subject Weight | Less than 1 minute
  Weight in kilograms
Collection of Subject Age | Less than 1 minute
  Age in years
Collection of Subject Medical Comorbidities | 1 minute
Systolic and Diastolic Blood Pressure Measurement | 1-2 minutes
  Using blood pressure cuff; measured three times to find the initial, interim, and final blood pressure
Collection of ECG Waveforms | 5 minutes
  Using an electrocardiogram (ECG) to measure heart rhythm
Collection of PPG Waveforms | 5 minutes
  Using a photoplethysmography (PPG) to monitor heart rate